CLINICAL TRIAL: NCT04642547
Title: A Prospective Clinical Study of Lenvatinib Combined With Gefitinib in the Treatment of Lenvatinib-resistant Hepatocellular Carcinoma
Brief Title: Lenvatinib Combined With Gefitinib in the Treatment of Lenvatinib-resistant Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhai Bo, Interventional Oncology Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJZLJRZB
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma; Molecular Targeted Therapy
Keywords: hepatocellular carcinoma; lenvatinib; gefitinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy with Lenvatinib and Gefitinib (Experimental): First week: Gefitinib 125mg/day, Lenvatinib 8mg/day if body weight ≤ 60Kg and 12mg/day if body weight > 60Kg. If the patient is well tolerated, the dose of Gefitinib will be adjusted to 250 mg/day after one week, and the dose of Lenvatinib will remain the same (8mg/day for weight ≤ 60Kg and 12mg/day for weight > 60Kg). Route of administration: Oral.
  Interventions: Drug: Lenvatinib and Gefitinib

INTERVENTIONS:
Drug: Lenvatinib and Gefitinib — First week: Gefitinib: 125mg/day, oral; Lenvatinib: 8mg/day (weight ≤ 60Kg) or 12mg/day (weight > 60Kg), oral.
  One week later: Gefitinib: 250mg/day, oral; Lenvatinib: 8mg/day (weight ≤ 60Kg) or 12mg/day (weight > 60Kg), oral.

SUMMARY:
This is a prospective clinical study aiming to tests the safety and efficacy of lenvatinib in combination with gefitinib in people with lenvatinib resistant hepatocellular carcinoma. This study will help find out if lenvatinib and gefitinib is a safe and useful combination for treating patients with lenvatinib resistant hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

(1) Unlimited gender, aged 18-75 years; (2) Meets American Association for the Study of Liver Diseases (AASLD) or European Association for the Study of the Liver (EASL) clinical diagnostic criteria of hepatocellular carcinoma; (3) Barcelona Clinic Liver Cancer (BCLC) Stage B or C, and there is at least one measurable tumor in the liver (long diameter ≥ 1cm);(4) progressing after standard treatment; (5) Unresponsive or resistant to Lenvatinib; (6) Child-Pugh A or scored 7 B; (7) Eastern Cooperative Oncology Group performance status score <= 1; (8) Platelet count >= 60x10^9/L, Prothrombin time prolonged <= 6 seconds.

Exclusion Criteria:

(1) Uncorrectable coagulopathy with obvious bleeding tendency; (2) Patients need long-term anticoagulant or anti platelet therapy and cannot stop the drugs; (3) Patients with unstable or active ulcer or gastrointestinal bleeding; (4) Heart disease requiring treatment or not well controlled high blood pressure; (5) Patients with interstitial pneumonia; (6) Hepatic encephalopathy or refractory ascites requiring treatment; (7) There is a clear active infection; (8) Receiving radiotherapy/chemotherapy/interventional therapy for tumor within 4 weeks before the start of the study; (9) Severe insufficiency of important organs, such as severe cardiopulmonary insufficiency; (10) Other accompanying anti-tumor treatments; (11) The investigator assessed that the patient was unable or unwilling to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 months after the last subject is enrolled
  The estimation of time from start of combination therapy to progression of disease

SECONDARY OUTCOMES:
Overall survival | 6 months after the last subject is enrolled
  The time between initial combination therapy and the patient's death of any cause or most recent follow-up.
Safety endpoint | 6 months after the last subject is enrolled
  Statistically describe the proportion of adverse events after treatment for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhai, MD&PhD, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shi Y, Cui D, Xia L, Shi D, Jin G, Wang S, Lin Y, Tang X, Chi J, Wang T, Li M, Lv Z, Zheng J, Jia Q, Yang W, Sun Z, Yang F, Feng H, Yuan S, Zhou W, Qin W, Bernards R, Jin H, Zhai B. Efficacy and safety of lenvatinib plus gefitinib in lenvatinib-resistant hepatocellular carcinomas: a prospective, single-arm exploratory trial. Signal Transduct Target Ther. 2024 Dec 9;9(1):359. doi: 10.1038/s41392-024-02085-8. PMID 39653700
- [Derived] Jin H, Shi Y, Lv Y, Yuan S, Ramirez CFA, Lieftink C, Wang L, Wang S, Wang C, Dias MH, Jochems F, Yang Y, Bosma A, Hijmans EM, de Groot MHP, Vegna S, Cui D, Zhou Y, Ling J, Wang H, Guo Y, Zheng X, Isima N, Wu H, Sun C, Beijersbergen RL, Akkari L, Zhou W, Zhai B, Qin W, Bernards R. EGFR activation limits the response of liver cancer to lenvatinib. Nature. 2021 Jul;595(7869):730-734. doi: 10.1038/s41586-021-03741-7. Epub 2021 Jul 21. PMID 34290403